CLINICAL TRIAL: NCT05784454
Title: Prevalence of Sleep Bruxism in a Group of Egyptian Children and Its Relation to Screen Time and Sugar Consumption
Brief Title: Prevalance of Sleep Bruxism Among a Group of Egyptian Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mira Ashraf Kamal, Doctor, Cairo University
Other Study IDs: Sleep Bruxism in Children
Record Dates: First submitted 2023-03-05; First posted 2023-03-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Sleep Bruxism
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this observational study is to detect the prevalence of sleep bruxism in a group of Egyptian children and detect its relation to screen-time and sugar consumption. The main questions it aims to answer are:

1. In a group of Egyptian Children what is the prevalence of sleep bruxism?
2. What is the relation between sleep bruxism and screen time and sugar consumption?

DETAILED DESCRIPTION:
Parents of a group of Egyptian Children aged 6-8 years old will be asked to fill

1. An informed Consent
2. Children Sleep Habit Questionnaire to detect the presence of sleep bruxism or not?
3. Food Frequency Questionnaire of Health Behaviour Sugar Consumption questionnaire
4. Leisure Time, Television Use, Computer Use Sections of the Health Behaviour Sugar Consumption Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Positive Subject acceptance for participation in the study
* Healthy children aged 6-8 years old
* Both genders
* The presence of mixed dentition with permnant first molar erupted

Exclusion Criteria:

* Children with mental or neurological disorders
* Children with systemic disorders
* Children who use medications that could not interfere with the central nervous system
* Children suffering from sleep disorders. e.g: Obstructive Sleep Apnea

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be selected according to the mentioned eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 349 (Estimated)
Dates: Start 2023-05-02 (Estimated); Primary Completion 2023-09-02 (Estimated); Study Completion 2023-11-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Sleep Bruxism in a group of Egyptian Children aged 6-8 years old | 1 year
  Cross sectional Observational Study

SECONDARY OUTCOMES:
Correlation between sleep bruxism and screen time and sugar consumption | 1 year
  Cross sectional Observational Study

CONTACTS AND LOCATIONS:
Overall Officials: Mira A Kamal, Bachelor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Restrepo C, Santamaria A, Manrique R. Sleep bruxism in children: relationship with screen-time and sugar consumption. Sleep Med X. 2021 Apr 24;3:100035. doi: 10.1016/j.sleepx.2021.100035. eCollection 2021 Dec. PMID 34169271
- See also: The link is to a similar article but with different age groups and different setting place — https://pubmed.ncbi.nlm.nih.gov/34169271/